CLINICAL TRIAL: NCT03613623
Title: Acromegaly: Patient And Physician Perspectives
Status: Completed | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: Chiasma, Inc. (Industry)
Responsible Party: Principal Investigator, Lizheng Shi, Principal Investigator, Tulane University
Other Study IDs: 2018-879
Record Dates: First submitted 2018-07-02; First posted 2018-08-03 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients diagnosed with acromegaly and currently taking long-acting somatostatin analogues for treatment.
- Physicians: Physicians for those treating the patients enrolled in the study.

SUMMARY:
The purpose of the study is to assess the experiences of individuals with acromegaly who are receiving injections as part of their treatment regimen. Another objective of the study is to compare the patients' perception with their doctors' perceptions. The answers are important to help researchers and physicians understand what it is really like to take currently available treatments so that they can make efforts to improve patients' healthcare experiences, reduce treatment burden and, ultimately, improve patient's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years-old and <95 years-old
* Patient self-reported acromegaly diagnosis which will be further confirmed by a knowledge screening based on current medications and doses
* Currently on injectable Somatostatin analogues (SSA), Sandostatin® LAR or Somatuline® Depot, for >=12 months
* Have not had a change in dosage of their acromegaly treatment at the time of or since their last office visit
* Have seen their treating acromegaly physician within the past 12 +/-2 months NOTE: This timeframe allows two additional months for scheduling an appointment with their physician, since most patients should see their acromegaly physician at least once every 12 months
* Ability to read and understand English
* Live and receive acromegaly treatments in the US
* Willing to provide signed informed consent

Exclusion Criteria:

* Previous or current participant in Mycapssa® (octreotide capsules) trial
* Use of Pegvisomant (Somavert®) monotherapy
* Use of Pasireotide (Signifor®)

Ages: 18 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acromegaly will be sent invitations to participate. Their physicians will be identified at the time of participant enrollment and will be contacted by the study team for a telephone interview.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Assess patient experiences with acromegaly treatments through patient questionnaires. | The questionnaire should take no more than 60 minutes per subject.
  The primary objective of this study is to assess the experience of patients treated with SSA injections in the United States. Patients will be asked about previous and current acromegaly treatments they have taken from the time of diagnosis to the current day they are completing the survey.
Assess patient satisfaction with acromegaly treatments. | The questionnaire should take no more than 60 minutes per subject.
  The primary objective of this study is to assess the treatment satisfaction of patients treated with SSA injections in the United States. Patients will be asked about previous and current acromegaly treatments they have taken from the time of diagnosis to the current day they are completing the survey.
Assess patients with acromegaly health-related quality of life. | The questionnaire should take no more than 60 minutes per subject.
  The primary objective of this study is to assess the health-related quality of life for patients treated with SSA injections in the United States. Patients will be asked about their current quality of life and how acromegaly and acromegaly treatments may affect their quality of life from time of diagnosis to time of completing the survey.

SECONDARY OUTCOMES:
Assess the concordance between patient's and physician's perceptions of acromegaly control (with/without biochemical lab results), | The questionnaire should take no more than 60 minutes per subject.
  The second objective of this study is to compare patients' perception with those of their physicians in terms of aspects such as acromegaly control, treatment satisfaction, and health-related quality of life (HRQoL).
Assess the concordance between patient's and physician's perceptions of acromegaly treatment satisfaction. | The questionnaire should take no more than 60 minutes per subject.
  The second objective of this study is to compare patients' perception with those of their physicians in terms of aspects such as acromegaly treatment satisfaction.
Assess the concordance between patient's and physician's perceptions of health-related quality of life. | The questionnaire should take no more than 60 minutes per subject.
  The second objective of this study is to compare patients' perception with those of their physicians in terms of aspects such as health-related quality of life (HRQoL).

CONTACTS AND LOCATIONS:
Overall Officials: Lizheng Shi, PhD, MsPharm, Principal Investigator — Tulane University
Locations (1):
- Tulane School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided